CLINICAL TRIAL: NCT03874845
Title: Neural Mechanisms of Mindfulness-based Cognitive Therapy (MBCT) for Posttraumatic Stress Disorder (PTSD)_single Site
Brief Title: Neural Mechanisms of Mindfulness-based Cognitive Therapy (MBCT) for Posttraumatic Stress Disorder (PTSD)_VA Only
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study had IRB approval from VA and began in late Feb 2020, did not enroll any participants before paused during the COVID. Final permissions from VA to restart recruitment was never received and therefore was withdrawn.
Sponsor: Ohio State University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Anthony P King, Associate Professor of Psychiatry, Faculty Associate, Institute for Behavioral Medicine Research, Institute for Behavioral Medicine Research, Institute for Social Research, Ohio State University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HUM00152509.K23; K23MH112852 (NIH)
Record Dates: First submitted 2019-03-12; First posted 2019-03-14 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Post Traumatic Stress Disorder
Keywords: Mindfulness-Based Cognitive Therapy; Muscle Relaxation; fMRI; Group Psychotherapy
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Mindfulness-Based Cognitive Therapy

STUDY DESIGN:
Intervention Model Description: treatment groups will consist of a minimum of 4 participants (preferably 5-8). The statistician will randomize the groups once a sufficient number of participants have enrolled to ensure desired group size.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Statistician will not know the group assignment until blind is broken. Statistician randomizes the groups. Principal investigator will not know group assignment until blind is broken.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness-Based Cognitive Therapy (Experimental): Participants will have 8 weeks of group therapy and will be asked to do MBCT exercises for approximately 20-30 minutes on 5 or more days/week.
  Interventions: Behavioral: Mindfulness-Based Cognitive Therapy
- Muscle Relaxation Therapy (MRG) (Active Comparator): Participants will have 8 weeks of group therapy participants and will be asked to do MRG exercises for approximately 20-30 minutes on 5 or more days/week.
  Interventions: Behavioral: Muscle Relaxation Therapy

INTERVENTIONS:
Behavioral: Mindfulness-Based Cognitive Therapy — Participants will attend 8 weekly group therapy sessions. Prior to and after therapy participants will have assessments related to their PTSD, fill out surveys, and have an fMRI.
  Arms: Mindfulness-Based Cognitive Therapy
Behavioral: Muscle Relaxation Therapy — Participants will attend 8 weekly group therapy sessions. Prior to and after therapy participants will have assessments related to their PTSD, fill out surveys, and have an fMRI.
  Arms: Muscle Relaxation Therapy (MRG)

SUMMARY:
This study will examine the effects of psychotherapy as treatment for PTSD. This research will see how brain activity and brain connectivity is affected by Mindfulness Based Cognitive Therapy (MBCT) and Muscle Relaxation Therapy (MRT). Participants that qualify to be in this study will receive 8 weeks of group therapy in MBCT or MRT. Prior to receiving therapy participants will: complete baseline assessments related to their PTSD; fill out surveys; have an functional magnetic resonance imaging (fMRI); and provide a saliva sample. These assessments will be repeated after the therapy is over. Overall study participation should last approximately 10-12 weeks.

DETAILED DESCRIPTION:
Note: due to COVID precautions, treatment shifted from in-person to remote ("Zoom" videoconferencing)

ELIGIBILITY:
Inclusion Criteria:

* Meets current Diagnostic and Statistical Manual of Mental Disorders, fifth edition (DSM-5) criteria for PTSD (with or without Major Depressive Disorder) or subsyndromal PTSD (qualifying trauma, and at least one intrusive, one avoidant, one negativity, and one arousal symptoms, and significant impairment or distress); type of trauma shall include interpersonal violence - combat, physical assault, sexual assault, etc.

Exclusion Criteria:

* Dissociative PTSD
* Delayed-onset PTSD
* Magnetic Resonance Imaging (MRI) contraindications (e.g. metal in body, inability to be in the scanner - claustrophobia, severe back pain, etc.)
* Serious medical or neurologic conditions (e.g. stroke, seizures)
* Suicide risk
* Psychosis
* Life history of schizophrenia
* Life history of bipolar disorder
* Current severe substance use disorder
* Other factors that preclude safe and meaningful participation in the study, at discretion of the PI and study team

Ages: 18 Years to 72 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-01-29 (Actual); Primary Completion 2023-03-30 (Estimated); Study Completion 2023-06-01 (Actual)

PRIMARY OUTCOMES:
Group differences in the change in resting-state functional connectivity between two large-scale distributed functional connectivity networks: the Default Mode Network (DMN) and the Central Executive Network (CEN) | pre-therapy and post therapy (approximately 8 weeks)
  Network functional connectivity will be measured through fMRI blood oxygen level dependent [BOLD] signal. Time-course of BOLD signal while participants are "resting" (not performing a task) will be used to identify patterns of functional connectivity between two large-scale neural networks DMN and CEN. We will use the Brain Basis Set methodology: creating a whole-brain correlation matrix between all combinations of hundreds of brain regions throughout the brain (a "connectome") followed by data-reduction methods (principle components analyses, PCA) to examine the structure of functional connectivity patterns between nodes of canonical intrinsic connectivity networks.

SECONDARY OUTCOMES:
Group differences in the change in resting-state functional connectivity between two large-scale distributed functional connectivity networks: the Default Mode Network (DMN) and the Salience Network (SN), measured through fMRI BOLD signal. | pre-therapy and post therapy (approximately 8 weeks)
  Network functional connectivity will be measured through fMRI blood oxygen level dependent [BOLD] signal. Time-course of BOLD signal while participants are "resting" (not performing a task) will be used identify patterns of functional connectivity between two large-scale neural networks DMN and CEN using the Brain Basis Set methodology.

CONTACTS AND LOCATIONS:
Overall Officials: Anthony King, Ph.D, Principal Investigator — University of Michigan and The Ohio State University
Locations (2):
- United States (2):
  - VA Ann Arbor Healthcare System, Ann Arbor, Michigan
  - The Ohio State University, Columbus, Ohio

IPD SHARING:
Plan to Share IPD: Yes
We plan to make available data from fMRI scans from human subjects initially to collaborators for independent replication / data pooling. We also plan to make the de-identified brain scans available to the broad scientific community, however, additional redaction steps may need to be made to brain scans to ensure subject confidentiality / inability to identify individuals from brain scans. Completely de-identified research data (redacted according to NIH practice to prevent disclosure of personal identifiers) which documents the research findings will be made available after the main findings from the finalized research dataset have been accepted for publication. And with approval of Dept Veterans Affairs Office of Research and Development.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Within 36 months of completion of the project.
Access Criteria: Access to data generated by the project will be available for educational, research and non-profit purposes to researchers who provide a methodologically sound proposal. Data generated under this project will be administered in accordance with NIH Sharing policies, including NIH Policy on Dissemination of NIH-Funded Clinical Trial Information (8/2016), and the NIH Grants Policy Statement (Availability of Research Results) (11/2015). Depending on such NIH policies, Data generated by this project may be available for educational, research or non-commercial purposes under the terms of a data use agreement. Data will be stored in an established data repository (e.g. Inter-university Consortium for Political and Social Research (ICPSR): icpsr.umich.edu) with appropriate provisions for curation and longterm preservation.